CLINICAL TRIAL: NCT04218227
Title: Dropout Factors in Chronic Pain Management : What Are the Predictors ?
Brief Title: Dropout Factors in Chronic Pain Management
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Audrey Vanhaudenhuyse, Principal Investigator, University of Liege
Other Study IDs: 2015/85-C
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Self Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Self-hypnosis/self-care group: It is a 7-months 2 hours-session (1 session per month) of self-hypnosis/self-care learning. Participants are given strategies to learn self-care (knowing their needs, self-respect, communication etc.), each strategy is discussed for participant to understand them and thus apply them correctly in daily life. An hypnosis exercice is conducted at the end of each session. A CD with the audiotaped hypnosis exercice is given to each patient so that they can practice also every day.
  Interventions: Behavioral: Self-hypnosis/self-care group
- Music/self-care: It is a 7-months 2 hours-session (1 session per month) of music/self-care learning. Participants are given strategies to learn self-care (knowing their needs, self-respect, communication etc.), each strategy is discussed for participant to understand them and thus apply them correctly in daily life. At the end of each session, patients are invited to listen to a relaxing melody of 15 minutes. This melody was composed by a professional musico-therapist. A CD with the audiotaped melody is given to each patient so that they can practice also every day.
  Interventions: Behavioral: Music/self-care
- Self-care: It is a 7-months 2 hours-session (1 session per month) of music/self-care learning. Participants are given strategies to learn self-care (knowing their needs, self-respect, communication etc.), each strategy is discussed for participant to understand them and thus apply them correctly in daily life.
  Interventions: Behavioral: Self-care
- Psycho-education: It is a 7-months 2 hours-session (1 session per month) of psycho-education training. Psycho-education aims to empower and encourage the patient to become an actor in his therapeutic management, while offering a comprehensive model of the mechanisms of pain, the benefits of pharmacological treatments at a physical and psychological level as well as ways to change the way one lives every day.
  Interventions: Behavioral: Psycho-education
- Self-hypnosis/self-care motivation: It is a 7-months 2 hours-session (1 session per month) of self-hypnosis/self-care learning. Participants are given strategies to learn self-care (knowing their needs, self-respect, communication etc.), each strategy is discussed for participant to understand them and thus apply them correctly in daily life. An hypnosis exercice is conducted at the end of each session. A CD with the audiotaped hypnosis exercice is given to each patient so that they can practice also every day.
  Interventions: Behavioral: Self-hypnosis/self-care motivation

INTERVENTIONS:
Behavioral: Self-hypnosis/self-care group — Self-hypnosis/self-care
  Groups: Self-hypnosis/self-care group
Behavioral: Music/self-care — Music-therapy/self-care
  Groups: Music/self-care
Behavioral: Self-care — Self-care
  Groups: Self-care
Behavioral: Psycho-education — Psycho-education
  Groups: Psycho-education
Behavioral: Self-hypnosis/self-care motivation — Motivation to learn self-hypnosis/self-care
  Groups: Self-hypnosis/self-care motivation

SUMMARY:
Chronic pain concernes one in four adults in Belgium. Because of the psychological and social repercussions, a biopsychosocial approach is necessary in order to improve the quality of life chronic pain patients. Non-pharmacological techniques such as hypnosis, self-care learning, music-therapy and psycho-education are gaining more and more interest in the scientific field. However, a major problem in clinical research is patient dropout. To our knowledge, no study has investigated dropout rates in hypnosis clinical research. The aim of this study is, therefore, to better understand the predictors of dropout in several non-pharmacological treatments in chronic pain management.

ELIGIBILITY:
Inclusion Criteria:

* Major
* Fluency in French
* Chronic pain diagnosis

Exclusion Criteria:

* Neurologic disorder
* Psychiatric disorder
* Drug addiction
* Alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have had a chronic pain diagnosis (all body-parts and all type of pain included) and must have been included in one of the outpatient chronic pain non-pharmacological management programme with an interdisciplinary approach proper to our pain department at the Hospital University of Liège (Belgium).
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Amount of drop-out | T1 (before treatment)
  The amount of drop-out between treatments group will be assessed by means of our database.
Amount of dropout between treatment groups | T1 (before treatment)
  The amount of drop-out between treatments group will be assessed by means of our database.
Influence of therapist's expertise in hypnosis | T1 (before treatment)
  The influence of the therapist's expertise in hypnosis upon drop-out will be assessed by means of our database.
Link between state-financial help and drop-out | T1 (before treatment)
  In Belgium, in certain cases, state will financially help patients to benefit from pain non-pharmacological treatments. We would like to understand if the benefit of state financial help influences the amount of drop-out.
Influence of motivation | T1 (before treatment)
  To understand of motivation influenced the amount of drop-out, we analysed the amount of drop-out in the "self-hypnosis/self-care motivation" group.
Influence of pain description | T1 (before treatment)
  The influence of pain description upon dropout rates will be assessed by means of a Visual Analogue Scale (VAS). Scale ranging from 0 (no pain) to 10 (worst pain).
Influence of sleep difficulties | T1 (before treatment)
  The influence of sleep difficulties upon dropout rates will be assessed by means of a Visual Analogue Scale (VAS). Scale ranging from 0 (no sleep difficulties) to 10 (worst sleep difficulties).
Influence of insomnia | T1 (before treatment)
  The influence of the severity of insomnia upon dropout will be assessed by means of the "Insomnia Severity Index" (Morin et al., 2001). Scale ranging from 0 (none) to 4 (very severe).
Influence of anxiety | T1 (before treatment)
  The influence of anxiety upon dropout will be assessed by means of the subtest "anxiety" of the Hospital Anxiety and Depression Scale (HADS, Zigmond & Snaith, 1983). Scale ranging from 0 (never) to 4 (always).
Influence of depression | T1 (before treatment)
  The influence of depression upon dropout will be assessed by means of the subtest "anxiety" of the Hospital Anxiety and Depression Scale (HADS, Zigmond & Snaith, 1983). Scale ranging from 0 (never) to 4 (always).
Influence of pain disability | T1 (before treatment)
  The influence of pain disability upon will be assessed by means of the "Pain Disability Index" (PDI, Tait et al., 1990). Scale ranging from 0 (no difficulties) to 10 (a lot of difficulties).
Influence of the impact of pain | T1 (before treatment)
  The influence of the impact of pain in individual's life, quality of social support and general activity, upon dropout will be assessed my means of the "Multidimensional Pain Index" (MPI, Kerns et al., 1985). Scale ranging from 0 (none) to 6 (a lot).
Influence of attitudes and beliefs about pain | T1 (before treatment)
  The influence of the attitudes and beliefs about pain upon dropout will be assessed my means of the "Survey of Pain Attitudes" (SOPA, Jensen & Karoly, 1987). Scale ranging from 0 (totally wrong) to 10 (totally right).
Influence of quality of life | T1 (before treatment)
  The influence of quality of life upon dropout will be assessed by means of the "SF-36"(Ware et al., 1988). Each item is balanced to obtain a score between 0 (worst quality) to 100 (maximum quality).
Influence of locus of control | T1 (before treatment)
  The influence of the locus of control upon dropoout will be assessd my means og the "Multidimensional Health Locus of Control" (MHLC, Wallston et al., 1978). Scale ranging from 1 (no agreement) to 4 (agreement).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital University of Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No